CLINICAL TRIAL: NCT04437043
Title: A Multicenter Belgian Trial on Ventral Hernia Repair. UNITE Study Protocol Number: RB-UNITE-01
Brief Title: A Multicenter Belgian Trial of Ventral Hernia Repair (UNITE)
Acronym: RB-UNITE-01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Royal Belgian Society for Surgery (Unknown); Archer Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BC-06967
Record Dates: First submitted 2020-03-11; First posted 2020-06-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Ventral Hernia
Keywords: ventral hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, academic, prospective, interventional, multicenter study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laparoscopic ventral hernia repair with closure of the defect (Other): In laparoscopic intraperitoneal onlay mesh or IPOM repair, the mesh is inserted intra-abdominally and fixed to the peritoneum / abdominal wall. The general steps include safe entry into the peritoneum, insufflation and placement of the trocars to gain access and visibility (via laparoscope) of the defect. Careful adhesiolysis is performed, which is the removal of scar tissue connecting tissues and organs. The content of the hernia, which may include intestine and fatty tissue, is returned into the abdominal cavity. After closure of the hernia defect, a wide intraperitoneal mesh is fixed over the defect. Desufflation releases the gas from the abdomen. The trocars will be removed and the incisions are closed.
  Interventions: Other: quality of life questionnaires
- Open ventral hernia repair with closure of the defect (Other): An open retromuscular ventral hernia repair involves an incision through the abdominal wall. Adhesiolysis is performed and the content of the hernia is returned into the abdominal cavity. The posterior rectus sheath is separated from the rectus muscle and closed, which closes the abdominal cavity. The mesh is then placed behind the muscle and anterior to the re-approximated posterior rectus sheath. Preperitoneal mesh extension is allowed via transversus abdominis release (TAR). The anterior rectus sheath is closed over the mesh, which closes the hernia.
  Interventions: Other: quality of life questionnaires
- Robotic ventral hernia repair with closure of the defect (Other): A robotic retromuscular ventral hernia repair involves a similar separation of the layers of the abdominal wall, similar closure of the hernia defect and similar retromuscular mesh placement as for the open approach. Preperitoneal mesh extension is allowed via TAR. The da Vinci System is a robotic-assisted surgical device that allows the surgeon to place long, narrow instruments through small incisions in order to perform surgery from the inside of the abdominal cavity. Rather than one long incision with open repair, four to six small incisions are made along the outer part of the abdomen between the rib cage and the hip.
  Interventions: Other: quality of life questionnaires

INTERVENTIONS:
Other: quality of life questionnaires — pain will be recorded in rest and activity (VAS) and patients will complete the quality of life questionnaires (CCS, BIQ). Also, the intake of analgesic medication will be registered. A clinical examination is conducted to evaluate the occurrence of seroma and to evaluate recurrence, defined as a protrusion of the contents of the abdominal cavity or preperitoneal fat through the defect, which is no longer covered by the mesh.

SUMMARY:
Patients with incisional midline ventral hernias with a minimal width of 3 cm and a maximal width of 8 cm, treated according to the standard practice of the participating investigators.

Patients can be treated with the following ventral hernia repair approaches:

* Laparoscopic ventral hernia repair with closure of the defect (IPOM+)
* Open ventral hernia repair with closure of the defect (retromuscular repair)
* Robotic ventral hernia repair with closure of the defect (retromuscular repair)

To evaluate the total number of days spent in the hospital within a period of 90 days post-operative. This will be calculated by adding the hospital length of stay for initial surgery or index-procedure, length of stay for any additional readmission resulting from the surgery or re-interventions, and emergency room visits resulting from the surgery or Serious Adverse Event (SAE) related to the index-procedure.

Secondary objectives: To assess the safety, performance and efficacy of laparoscopic, open and robotic ventral hernia repair.

DETAILED DESCRIPTION:
Ventral hernia repair

1. Laparoscopic: In laparoscopic intraperitoneal onlay mesh or IPOM repair, the mesh is inserted intra-abdominally and fixed to the peritoneum / abdominal wall. The general steps include safe entry into the peritoneum, insufflation and placement of the trocars to gain access and visibility (via laparoscope) of the defect. Careful adhesiolysis is performed, which is the removal of scar tissue connecting tissues and organs. The content of the hernia, which may include intestine and fatty tissue, is returned into the abdominal cavity. After closure of the hernia defect, a wide intraperitoneal mesh is fixed over the defect. Desufflation releases the gas from the abdomen. The trocars will be removed and the incisions are closed.
2. Open: An open retromuscular ventral hernia repair involves an incision through the abdominal wall. Adhesiolysis is performed and the content of the hernia is returned into the abdominal cavity. The posterior rectus sheath is separated from the rectus muscle and closed, which closes the abdominal cavity. The mesh is then placed behind the muscle and anterior to the re-approximated posterior rectus sheath. Preperitoneal mesh extension is allowed via transversus abdominis release (TAR). The anterior rectus sheath is closed over the mesh, which closes the hernia.
3. Robotic: A robotic retromuscular ventral hernia repair involves a similar separation of the layers of the abdominal wall, similar closure of the hernia defect and similar retromuscular mesh placement as for the open approach. Preperitoneal mesh extension is allowed via TAR. The da Vinci System is a robotic-assisted surgical device that allows the surgeon to place long, narrow instruments through small incisions in order to perform surgery from the inside of the abdominal cavity. Rather than one long incision with open repair, four to six small incisions are made along the outer part of the abdomen between the rib cage and the hip.

Classifications and questionnaires

1. European Hernia Society (EHS) classification: The EHS classification is a simple and reproducible system, developed to allow comparison of publications and future studies on primary and incisional abdominal wall hernias. The classification includes the localization of the hernia as well as the size of the hernia defect as decisive for the outcome. The EHS classification is to be filled in by the participating investigator following the patients CT scan.
2. Post-Anaesthetic Discharge Scoring System (PADSS): The Modified PADSS has proven to be an efficient system that guarantees safe discharge. PADSS is based on the assessment of 6 criteria: vital signs (including blood pressure, pulse, temperature and respiratory rate), ambulation, nausea / vomiting, pain, surgical bleeding and fluid intake / output. Each criterion is given a score from 0 to 2. Patients scoring ≥ 9 are considered fit for discharge, provided that the score for vital signs is not lower than 2 and that none of the other five criteria is 0, even if the total score reaches 9. PADSS scoring will be performed twice a day, in the morning and in the afternoon with minimally 9 hours in between. Same day discharge (on the day of hernia repair) is allowed as long as the required PADSS score is reached.
3. American Society of Anesthesiologists (ASA) Classification: The ASA physical status classification system was developed to offer clinicians a simple categorization of a patient's physiological status that can be helpful in predicting operative risk.
4. Visual Analog Scale (VAS): The VAS scoring system is frequently used as a reliable and valid measure of pain. It contains a 0 - 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain. The patient is asked to select the number on the scale that corresponds to the worst level of pain he / she experiences in rest and activity. The patient will be asked to bend over to score pain during activity. Pain is classified into mild (1 - 30 mm), moderate (31 - 60 mm) and severe (61 - 100 mm). Absence of pain is defined as VAS = 0.
5. Carolinas Comfort Scale (CSS): The CCS is a disease-specific, quality of life questionnaire developed for patients undergoing hernia repair with mesh. It is a 23-item questionnaire that measures the severity of pain, sensation and movement limitations from the mesh in eight categories. The CCS score is derived by adding the scores from each of the 23 items. The best possible score is 0 and the worst possible score is 115.
6. Body Image Questionnaire (BIQ): The BIQ is an ten-item questionnaire incorporating body image and cosmetic subscales. The body image scale measures patients' perception and satisfaction with their bodies after surgery, and it is calculated by reverse scoring and summing the responses to questions 1 through 5. It ranges from 5 to 20 with a higher number representing greater body image perception. The cosmetic scale assesses satisfaction with surgical scars and is calculated by simply summing responses to questions 6 through 8, for a score range of 3 to 24, with a higher score indicating greater cosmetic satisfaction. The last two items (9, 10) score self-confidence before and after surgery. The Baseline BIQ was generated to score body image perception and satisfaction at baseline and consists of 9 questions.
7. Seroma classification: Seroma is one of the most common complications after hernia repair. The seroma classification is used to describe the incidence of seroma after ventral hernia repair and was developed in order to unify criteria among surgeons when describing their experience. Originally developed for seroma classification after laparoscopic ventral hernia repair, it can also be used to describe the incidence of seroma after open ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with incisional midline ventral hernia (M2: epigastric, M3: umbilical, M4: infra-umbilical) with a minimal width of 3 cm and a maximum width of 8 cm. Multiple hernia defects (Swiss cheese) are allowed according to European Hernia Society (EHS) classification (Appendix 1).
2. Recurrences are only allowed to be included after former primary repair (suture repair without mesh).
3. Patients with ASA grade I to III.
4. Patient is at least 18 years old.
5. Patient must sign and date the informed consent form prior to treatment.
6. Patient is able to tolerate general anesthesia.

Exclusion Criteria:

1. Patient with a life expectancy of less than 2 years.
2. Patient is suspected of being unable to comply with the study protocol.
3. Patient is pregnant.
4. Patient needs acute surgery.
5. Patient is enrolled in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Total number of days in the hospital | 90 days post-operative
  This will be calculated by adding the hospital length of stay for initial surgery, length of stay for any additional readmission resulting from the surgery, and emergency room visits resulting from the surgery. This information will be collected up to 90 days after the surgery. The hospital length of stay for the initial surgery will be assessed using a Modified Post Anaesthetic Discharge Scoring System (PADSS)

SECONDARY OUTCOMES:
Intra-operative adverse events | index procedure, 30 days post-operative, and 90 days post-operative
  Definitions according to ICH-GCP E6 (R2)
Number of participants with Surgical Site Infection (SSI) | post-operative at 30 days, 1 year, and 2 years
  CDC definition
Number of participants with Surgical Site Occurence (SSO) | post-operative at 30 days, 1 year, and 2 years
  Hematoma, seroma, dehiscence, necrosis, non-healing wound found on abdominal exam
Operating time | index procedure
  Total operating time from incision to last stitch (in minutes)
Effective day of discharge | index procedure, and post-operative at 30 days
  Number of effective hospital stay after the index procedure
Conversion rate | index procedure
  Conversion rate for the laparoscopic and robot-assisted groups
Preoperative and post-operative pain | enrollment, post-operative at 30 days, 1 year, and 2 years
  Pain scoring using the Visual Analog Scale (VAS) The VAS scoring system is frequently used as a reliable and valid measure of pain. It contains a 0 - 100 grading scale with 0 equaling no pain and 100 equaling the worst conceivable pain. The patient is asked to select the number on the scale that corresponds to the worst level of pain he / she experiences in rest and activity. The patient will be asked to bend over to score pain during activity. Pain is classified into mild (1 - 30 mm), moderate (31 - 60 mm) and severe (61 - 100 mm). Absence of pain is defined as VAS = 0.
Analgesic intake | post-operative at 30 days, 1 year, and 2 years
  Amount and type of analgesic intake
Quality of life improvement: Carolina's Comfort Scale (CCS) | enrollment, post-operative at 30 days, 1 year, and 2 years
  Carolina's Comfort Scale (CCS)
Body image | enrollment, post-operative at 30 days, 1 year, and 2 years
  Body Image Questionnaire (BIQ) The BIQ is a ten-item questionnaire incorporating body image and cosmetic subscales. The body image scale measures patients' perception and satisfaction with their bodies after surgery, and it is calculated by reverse scoring and summing the responses to questions 1 through 5. It ranges from 5 to 20 with a higher number representing greater body image perception. The cosmetic scale assesses satisfaction with surgical scars and is calculated by simply summing responses to questions 6 through 8, for a score range of 3 to 24, with a higher score indicating greater cosmetic satisfaction. The last two items (9, 10) score self-confidence before and after surgery.
Recurrence | post-operative at 30 days, 1 year, and 2 years
  Recurrent hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No